CLINICAL TRIAL: NCT03757767
Title: The Fasting Study - Unraveling the Mechanistic Effects of Prolonged Fasting in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lydia A. Afman, Principal Investigator, Wageningen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL-66589.081.18
Record Dates: First submitted 2018-11-09; First posted 2018-11-29 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Fasting; Adipose Tissue; Clinical Trial; Lipid Metabolism
Keywords: Physiology; Humans
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: Research subjects are measured in the fed state and in the prolonged fasted state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Fasting for 26-hours.
  Interventions: Other: Fasting for 26-hours

INTERVENTIONS:
Other: Fasting for 26-hours — All research subjects will have to fast for 26 hours in total.
  All research subjects start with a standardized meal. Two hours after the standardized meal the samples in the fed state will be taken. Research participants are not allowed to eat anything after the consumption of the standardized meal until the second measurements on day 2, 26-hours later. There are 24 hours between the two measurement points.
  Other Names: Prolonged fasting

SUMMARY:
Elevated levels of plasma triglycerides are increasingly recognized as an important causal risk factor for cardiovascular disease and associated pathologies. Lowering plasma triglycerides may therefore be a therapeutic target to lower cardiovascular disease risk. With this study the investigators want to examine the effects of fasting on adipose tissue metabolism in humans.

DETAILED DESCRIPTION:
Rationale: Elevated levels of plasma triglycerides are increasingly recognized as an important causal risk factor for cardiovascular disease and associated pathologies. Lowering plasma triglycerides may therefore be a therapeutic target to lower cardiovascular disease risk. Lipoprotein lipase (LPL) is the enzyme that catalyzes the hydrolysis of plasma triglycerides into fatty acids on the capillary endothelium, thereby lowering plasma triglycerides and stimulating the uptake of these fatty acids into cells. Angiopoietin-like 4 (ANGPTL4) is produced by fat cells and promotes the unfolding and inactivation of LPL, leading to decreased hydrolysis of plasma triglycerides. The role of ANGPTL4 in regulating LPL is especially important during fasting. However, as most studies are performed in animal models, little is known about the effects of fasting on adipose tissue metabolism in humans, and specifically on ANGPTL4 and its relationship with LPL.

Objectives: The key objective of this study is to determine the effect of a prolonged fast on ANGPTL4 gene and protein expression in subcutaneous adipose tissue, the key organ involved in lipid metabolism. Additionally, the effect of a prolonged fast on LPL gene expression, LPL protein expression, and on LPL activity in subcutaneous adipose tissue will be examined. To explore the systemic effects of a prolonged fast, the investigators will also measure ANGPTL4 levels in plasma, and ANGPTL4 and LPL gene expression in circulating immune cells (PBMCs). The secondary objective of this study is to obtain a more holistic view on the changes occurring upon a prolonged fast, by examining the effects of fasting on whole genome expression, post-transcriptional changes, and on markers of metabolic status. The combined results of all measurements will ultimately lead to a better understanding of the mechanistic effects of a prolonged fast and the metabolic functioning in humans.

Study design: The Fasting Study is a single arm intervention study in healthy men and women. The investigators will examine the effects of a fed state, which is 2 hours after the last food intake, versus a prolonged fasted state, which is 26 hours after the last food intake. Adipose tissue biopsies and blood samples will be taken 2 hours after the last meal and 26 hours after the last meal. The 24 hours between sampling points are chosen to prevent effects of the circadian rhythm.

Study population: The study population will consist of 24, 40-70 years old men and women with a BMI of 22-30 kg/m2, selected from the surroundings of Wageningen through the mailing list for potential study research subjects of the division of Human Nutrition and health of Wageningen University. If needed, additional recruitment of research subjects will take place by flyers and posters, or advertisements in local newspapers.

Intervention: All research subjects will start with the consumption of a standardized meal (ad libitum). Directly thereafter the intervention begins, which is a fasting period of twenty-six-hours, during which research subjects are not allowed to eat or drink anything except for water, which the research subjects may consume ad libitum. The investigators will take the first blood samples and adipose tissue biopsies two hours after the consumption of the standardized meal. This is the fed state: the point in time where the body is physiologically fed, based on the average time for plasma free fatty acids to drop. Twenty-four hours after the "fed state", research subjects are in the prolonged fasted state, and the investigators will take the final blood samples and adipose tissue biopsies. The time period of twenty-four-hours between sampling points is chosen to prevent the effects of circadian related changes on our outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy man or woman
* Age 40-70y at the time of recruitment
* BMI of 22-30 kg/m2
* Willing to fast for 26 hours
* Willing to give blood samples
* Willing to give adipose tissue biopsies
* Willing to consume the standardized meal on test day 1
* Signed informed consent
* Having a general practitioner

Exclusion Criteria:

* Alcohol on average: more than 2 consumptions/day or more than 14 consumptions/week
* Tobacco smoker
* Usage of drugs
* Following a diet within one month of starting the study (for example a ketogenic diet)
* Allergic to one or more components of the standardized meal
* Donated or intend to donate blood from 2 months before the study until the end of the study
* Unstable body weight (weight gain or loss >5 kg in the past three months)
* Diagnosed with any long-term medical condition that can interfere with the study outcome (i.e. cardiovascular disease, diabetes mellitus type 1 or 2, liver, pulmonary, or renal disease)
* Use of prescribed medication
* Use of supplements or over the counter medication (OTC) known to interfere with glucose or lipid homeostasis in the week before the start of the study, and during the study
* Being pregnant or lactating
* Participation in another biomedical study (other than the EetMeetWeet study) during this study
* Members of the research team, or first degree family members of the research team
* Working, or doing an internship at the division "Human Nutrition and Health" - Wageningen University

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Change in ANGPTL4 protein and gene expression in adipose tissue | there are 24 hours between the measurement in de fed and the fasted state
  Using Western blotting, the change in ANGPTL4 protein expression in adipose tissue will be measured from fed to a prolonged fasted state. The change in ANGPTL4 gene expression in adipose tissue will be measured from fed to a prolonged fasted state using whole genome affymetrix microarrays and targeted quantitative real time PCR.
Change in LPL expression, both gene and protein, and LPL activity in adipose tissue | There are 24 hours between the measurement in the fed and the fasted state
  Using Western blotting, the change in LPL protein expression in adipose tissue will be measured from fed to a prolonged fasted state. The change in LPL gene expression in adipose tissue will be measured from fed to a prolonged fasted state using whole genome affymetrix microarrays and targeted quantitative real time PCR. The change in LPL activity in subcutaneous adipose tissue will be measured from fed to a prolonged fasted state, using a lipoprotein lipase assay.
Change in ANGPTL4 expression in plasma | There are 24 hours between the measurement in the fed and the fasted state
  Using ELISA, the change in ANGPTL4 expression in plasma will be measured from fed to a prolonged fasted state.
Change in ANGPTL4 and LPL gene expression in PBMCs | There are 24 hours between the measurement in the fed and the fasted state
  The change in ANGPTL4 and LPL gene expression in PBMCs from fed to a prolonged fasted state will be measured using whole genome affymetrix microarrays and targeted quantitative real time PCR.

SECONDARY OUTCOMES:
Change in whole genome expression | There are 24 hours between the measurement in the fed and the fasted state
  Using whole genome affymetrix micorarrays, the change in whole genome gene expression in both adipose tissue and PBMCs will be measured from fed to a prolonged fasted state.
Post-transcriptional changes | There are 24 hours between the measurement in the fed and the fasted state
  Using microRNAarrays of Thermo Fisher Scientific, targeted digital droplet PCR, and quantitative real time PCR, post-transcriptional changes in adipose tissue and PBMCs will be measured from fed to a prolonged fasted state.
Changes in metabolite profiles | There are 24 hours between the measurement in the fed and the fasted state
  Using untargeted and targeted metabolomic platforms, the changes in metabolite profiles in the adipose tissue and plasma/serum will be measured.
Changes in protein profiles | There are 24 hours between the measurement in the fed and the fasted state
  Using untargeted and targeted proteomic platforms, the changes in protein profiles in the adipose tissue and plasma/serum will be measured.

OTHER OUTCOMES:
BMI | At baseline
  weight (in kg) and height (in meters) will be measured and combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Afman, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Collected data will be coded.

REFERENCES:
- [Derived] Ruppert PMM, Michielsen CCJR, Hazebroek EJ, Pirayesh A, Olivecrona G, Afman LA, Kersten S. Fasting induces ANGPTL4 and reduces LPL activity in human adipose tissue. Mol Metab. 2020 Oct;40:101033. doi: 10.1016/j.molmet.2020.101033. Epub 2020 Jun 3. PMID 32504883